CLINICAL TRIAL: NCT04409353
Title: Randomized-controlled Trial of Virtual Reality for Chronic Low Back Pain to Improve Patient-reported Outcomes and Physical Activity
Brief Title: Virtual Reality Therapy for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Brennan Spiegel, Staff Physician III, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00000631; 1UG3AR076573-01 (NIH)
Record Dates: First submitted 2020-05-14; First posted 2020-06-01 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low Back Pain
Keywords: Virtual Reality; Chronic Low Back Pain; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Providers, Primary Investigator, and Biostatistician were all blinded to allocations until the end of data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Distraction-Based VR (Active Comparator): EaseVRx-Distraction has the same number of experiences, the same approximate duration of experiences, and the identical user interface as EaseVRx+, with a linear prescribed sequence of experiences. The key differences are the lack of an on-demand library and that instead of offering a variety of VR experiences including education, games, and breath biofeedback, EaseVRx Distraction only includes 360-degree videos - which are also present in EaseVRx+. This is intended to remove the effect of education and skills-based training, while preserving the immersive experience of 360- degree VR.
  Interventions: Device: Distraction-Based VR; Device: Activity Tracker
- Sham VR (Sham Comparator): EaseVRx-Sham software includes 2D nature footage accompanied by neutral music that is selected to be neither relaxing nor distracting, rather than 360-degree, 3D, interactive content specially selected for efficacy. The experience of using EaseVRx-Sham is similar to watching a large-screen TV, but it is not interactive or immersive. EaseVRx Sham has the same number and duration of experiences as the EaseVRx+ linear prescribed sequence but does not contain an on-demand library; the functionality of the user interface used to access the experiences is otherwise the same as EaseVRx+. Modifications were made to the appearance of the user interface in order to remove aspects that were added for therapeutic benefit.
  Interventions: Device: Sham VR; Device: Activity Tracker
- Skills-Based VR (Experimental): EaseVRx+ incorporates the evidence-based principles of CBT, mindful meditation, and physiologic biofeedback therapy using embedded biometric sensors. It combines psychoeducation, pain education, breathing training, relaxation exercises, and executive functioning games to provide a mind-body approach toward living better with chronic pain. The standardized, prescriptive, and reproducible 56-day program delivers a combination of skills training and CBT-related treatments through scheduled daily virtual experiences. EaseVRx+ also features an on-demand library, allowing users to access any of the unique video sessions as needed.
  Interventions: Device: Skills-Based VR; Device: Activity Tracker

INTERVENTIONS:
Device: Distraction-Based VR — Participants will use the Pico G2 4K VR audio and visual head-mounted device, loaded with the EaseVRx-Distraction software. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view. The headset battery requires recharging after approximately 2.5 hours of use.
  https://www.pico-interactive.com/us/G2_4K.html
  Other Names: EaseVRx-Distraction Software; PICO G2 4k
  Arms: Distraction-Based VR
Device: Sham VR — Participants will use the Pico G2 4K VR audio and visual head-mounted device, loaded with the EaseVRx-Sham software. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view. The headset battery requires recharging after approximately 2.5 hours of use.
  https://www.pico-interactive.com/us/G2_4K.html
  Other Names: EaseVRx-Sham Software; PICO G2 4k
  Arms: Sham VR
Device: Skills-Based VR — Participants will use the Pico G2 4K VR audio and visual head-mounted device, loaded with the EaseVRx+ software. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view. The headset battery requires recharging after approximately 2.5 hours of use.
  https://www.pico-interactive.com/us/G2_4K.html
  Other Names: EaseVRx+ Software; PICO G2 4k
  Arms: Skills-Based VR
Device: Activity Tracker — Participants among all arms will be provided the option to passively wear a Fitbit Charge 4 throughout their 90-day study enrollment period. The Fitbit collects biometric data such as daily steps, heart rate, hours of sleep, stages of sleep, and sleep efficiency.
  Other Names: Fitbit Charge 4

SUMMARY:
This study will test the efficacy of an evidence-based virtual reality (VR) therapy program as a non-pharmacological supplement for the management of chronic lower back pain. Study participants will be randomized to receive one of three VR programs: Skills-Based VR, Distraction VR, or Sham VR. In addition to a VR headset, all participants will receive a Fitbit Charge 4 watch. Study devices will be delivered to the participant's home with instructions for use via FedEx; participants will receive remote technical support. They will be followed for 90 days and complete Patient Reported Outcome (PRO) questionnaires to assess functional status, pain levels, and use of pain medications (including opioids). Participants will also be asked to provide consent/authorization to access medical records from their treating facility.

DETAILED DESCRIPTION:
This is a randomized double-blind, placebo-controlled trial for individuals with chronic lower back pain. This study investigates the effect of at-home virtual reality (VR) pain reduction therapies on a set of outcome measures. The primary outcome is Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference version 8. This study will enroll 360 analyzable participants into one of three VR therapy groups. Data collection will occur at home via personal computer or smartphone (iPhone/android), with baseline data collected one week before the intervention is mailed to the patient. Participants will have the VR headset for 90 days. Patients are also sent Fitbit smartwatches to track physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide consent to participate in research
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, age 13 or older
4. An ongoing low back-pain problem that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months.
5. Ability to comprehend spoken and written English
6. Owns a compatible android or iOS smartphone, or personal laptop or desktop computer (excluding tablets) to complete surveys and has access to email.

Exclusion Criteria:

1. Presents with a condition that interferes with virtual reality usage, including history of seizure, facial injury precluding safe placement of headset, significant visual or hearing impairment that impacts ability to see the virtual reality images or follow audio instructions
2. Are being recommended for long-term hospitalization that would require more than three-week stay in the hospital
3. Received surgical procedure within the previous 8 weeks
4. Surgery is planned within the next 3 months
5. Is currently using a spinal cord stimulator
6. Has low back pain attributable to a recognizable, specific pathology, including spinal infection, cancer, fracture, or inflammatory spondylopathies, consistent with the NIH Task force on Research Standards for chronic low back pain
7. Previously participated in a virtual reality clinical trial

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, Principal Investigator — Cedars-Sinai
Locations (1):
- Samuel Eberlein, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
This study is part of the NIH Helping to End Addiction Long-term (HEAL) Initiative focused on understanding and developing new treatments for addiction and pain. Deidentified patient data, including demographics and longitudinal patient reported outcomes (PROs) are uploaded to the Back Pain Consortium (BACPAC) Data Portal.
Time Frame: 2020 to 2024
Access Criteria: The researcher must be part of the NIH Back Pain Consortium (BACPAC) consortium.
URL: https://www.bacpacresearch.org/

REFERENCES:
- [Derived] Birckhead B, Eberlein S, Alvarez G, Gale R, Dupuy T, Makaroff K, Fuller G, Liu X, Yu KS, Black JT, Ishimori M, Venuturupalli S, Tu J, Norris T, Tighiouart M, Ross L, McKelvey K, Vrahas M, Danovitch I, Spiegel B. Home-based virtual reality for chronic pain: protocol for an NIH-supported randomised-controlled trial. BMJ Open. 2021 Jun 15;11(6):e050545. doi: 10.1136/bmjopen-2021-050545. PMID 34130965
- See also: Study web portal for more information and a self-assessment for eligibility — https://virtualmedicine.org/research/current/vr4backpain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Cedars-Sinai physician partners at outpatient pain clinic, spine center, rheumatology, community partners such as the ACPA and Saban Clinic, and/or pulled directly from the medical record database between September 2020 and October 2023. All enrollment activities were conducted remotely, by telephone and electronic survey. Recruitment spanned from 10/21/2020 to 10/17/2023. 385 total participants were recruited, producing a final analyzable sample N=360.
Pre-assignment Details: Of 1,213 screened participants, 413 met inclusion criteria and signed an eConsent form. Of these, only 385 successfully completed the minimum required 4 of 7 screening week surveys and were randomized to treatment.
Groups:
- Distraction-Based VR: EaseVRx-Distraction has the same number of experiences, the same approximate duration of experiences, and the identical user interface as EaseVRx, with a linear prescribed sequence of experiences. The key difference is that instead of offering a variety of VR experiences including education, games, and breath biofeedback, EaseVRx Distraction only includes 360-degree videos - which are also present in EaseVRx. This is intended to remove the effect of education and skills-based training, while preserving the immersive experience of 360- degree VR.
  Distraction-Based VR: Participants will use the Pico G2 4K VR audio and visual head-mounted device, loaded with the EaseVRx-Distraction software. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view. The headset battery requires recharging after approximately 2.5 hours of use.
  https://www.pico-interactive.com/us/G2_4K.html
  Activity Tracker: Participants among all arms were given the option to passively wear a Fitbit Charge 4 throughout their 90-day study enrollment period. The Fitbit collected biometric data such as daily steps, heart rate, hours of sleep, stages of sleep, and sleep efficiency.
- Sham VR: EaseVRx-Sham software includes 2D nature footage accompanied by neutral music that is selected to be neither relaxing nor distracting, rather than 360-degree, 3D, interactive content specially selected for efficacy. The experience of using EaseVRx-Sham is similar to watching a large-screen TV, but it is not interactive or immersive. EaseVRx Sham has the same number and duration of experiences as EaseVRx, and the functionality of the user interface used to access the experiences is the same. Modifications were made to the appearance of the user interface in order to remove aspects that were added for therapeutic benefit.
  Sham VR: Participants will use the Pico G2 4K VR audio and visual head-mounted device, loaded with the EaseVRx-Sham software. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view. The headset battery requires recharging after approximately 2.5 hours of use.
  https://www.pico-interactive.com/us/G2_4K.html
  Activity Tracker: Participants among all arms were given the option to passively wear a Fitbit Charge 4 throughout their 90-day study enrollment period. The Fitbit collected biometric data such as daily steps, heart rate, hours of sleep, stages of sleep, and sleep efficiency.
- Skills-Based VR: EaseVRx+ incorporates the evidence-based principles of CBT, mindful meditation, and physiologic biofeedback therapy using embedded biometric sensors. It combines psychoeducation, pain education, breathing training, relaxation exercises, and executive functioning games to provide a mind-body approach toward living better with chronic pain. The standardized, prescriptive, and reproducible 56-day program delivers a combination of skills training and CBT-related treatments through scheduled daily virtual experiences. EaseVRx+ also features an on-demand library, allowing users to access any of the unique video sessions as needed.
  Skills-Based VR: Participants will use the Pico G2 4K VR audio and visual head-mounted device, loaded with the EaseVRx+ software. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view. The headset battery requires recharging after approximately 2.5 hours of use.
  https://www.pico-interactive.com/us/G2_4K.html
  Activity Tracker: Participants among all arms were given the option to passively wear a Fitbit Charge 4 throughout their 90-day study enrollment period. The Fitbit collected biometric data such as daily steps, heart rate, hours of sleep, stages of sleep, and sleep efficiency.
Period: Overall Study
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Started | 127 | 127 | 131
Follow-Up Complete (Completed survey follow-up - may have discontinued use of intervention) | 107 | 111 | 111
Completed (Completed protocol (follow-up complete and did not discontinue intervention)) | 103 | 100 | 105
Not Completed | 24 | 27 | 26
Not completed — Discontinued intervention prior to end of follow-up | 4 | 11 | 6
Not completed — Lost to Follow-up | 6 | 8 | 7
Not completed — Major surgery during participation window | 4 | 3 | 3
Not completed — Life event occurred during participation window | 3 | 2 | 4
Not completed — Lack of Efficacy | 4 | 1 | 3
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Disease burden - unable to participate | 0 | 1 | 1
Not completed — Intervention too complicated | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR | Total
Number analyzed (Participants) | 127 | 127 | 131 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (14.6) | 52.4 (16.5) | 54.8 (15.7) | 54.1 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 81 | 86 | 241
  Male | 53 | 46 | 45 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 30 | 31 | 93
  Not Hispanic or Latino | 93 | 93 | 95 | 281
  Unknown or Not Reported | 2 | 4 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 | 4
  Asian | 8 | 7 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 25 | 29 | 21 | 75
  White | 85 | 77 | 89 | 251
  More than one race | 2 | 3 | 6 | 11
  Unknown or Not Reported | 7 | 8 | 10 | 25
Education [Count of Participants; unit: Participants]
  Upper Secondary (High School) | 2 | 2 | 3 | 7
  High School diploma or equivalent (GED) | 8 | 6 | 7 | 21
  Some College/Certificate | 30 | 28 | 35 | 93
  Vocational/Trade School | 10 | 9 | 9 | 28
  Bachelor's Degree | 37 | 36 | 31 | 104
  Some Graduate School or Professional School | 8 | 9 | 11 | 28
  Graduate or Professional School diploma | 32 | 37 | 35 | 104
Employment [Count of Participants; unit: Participants]
  Full-time employment | 41 | 53 | 38 | 132
  Not employed | 25 | 20 | 36 | 81
  Part-time employment | 18 | 17 | 16 | 51
  Retired | 43 | 37 | 41 | 121
Marital Status [Count of Participants; unit: Participants]
  Divorced | 19 | 19 | 17 | 55
  Married | 46 | 59 | 57 | 162
  Never married | 40 | 34 | 43 | 117
  Separated | 2 | 1 | 1 | 4
  Widowed | 11 | 6 | 6 | 23
  Domestic Partner | 9 | 8 | 7 | 24
Income [Count of Participants; unit: Participants]
  Less than $10,000 | 6 | 7 | 9 | 22
  $10,000-$24,999 | 17 | 10 | 20 | 47
  $25,000-$34,999 | 13 | 5 | 3 | 21
  $35,000-$49,999 | 11 | 9 | 14 | 34
  $50,000-$74,999 | 16 | 18 | 15 | 49
  $75,000-$99,999 | 16 | 16 | 14 | 46
  $100,000-$149,999 | 14 | 21 | 18 | 53
  $150,000-$199,999 | 9 | 8 | 8 | 25
  $200,000 or more | 12 | 16 | 10 | 38
  Prefer not to answer | 13 | 17 | 20 | 50
Average of daily back pain assessments [Mean (Standard Deviation); unit: units on a scale] — Baseline measure refers to the average of daily assessments for self-reported back pain on an 11-point scale from 0 (No Pain) to 10 (Pain as bad as you can imagine) over a 7-day screener week for 385 participants. Participants were asked to report their pain scores each day for the. Each participant provided at least 4 of the 7 assessments to qualify for the study. The average of all available measurements for each participant was computed, then averages of averages were computed by arm. Higher scores indicate worse pain.
  units on a scale | 6.0 (1.9) | 6.0 (1.9) | 6.3 (1.9) | 6.1 (1.9)
Average low-back pain in past 7 days [Mean (Standard Deviation); unit: units on a scale] — Baseline measure refers to the average self-reported back pain on an 11-point scale from 0 (No Pain) to 10 (Pain as bad as you can imagine) for 385 participants. Participants were asked to recall and report their average back pain in the past 7 days during a single measurement during the 7-day screener week. Averages were computed by arm. Higher scores indicate worse pain.
  units on a scale | 5.8 (1.9) | 5.8 (1.8) | 5.9 (2.0) | 5.8 (1.9)
Opioid Use [Count of Participants; unit: Participants] — Measure of the number of participants who self-report opioid use at the start of the trial, collected during 7-day screener week prior to randomization.
  Participants
    Yes | 41 | 36 | 40 | 117
    No | 84 | 90 | 89 | 263
    Not sure | 2 | 1 | 2 | 5
Back Pain Severity [Count of Participants; unit: Participants] — Measure of the number of participants who self-reported that their lower back pain was more severe than pain in other parts of their body. Collected during 7-day screener week prior to randomization.
  Participants
    Yes | 92 | 94 | 96 | 282
    No | 20 | 21 | 20 | 61
    Not sure | 15 | 12 | 15 | 42
Back Pain Operation [Count of Participants; unit: Participants] — Measure of the number of participants who self-reported their previous surgical history for their lower back. Collected during 7-day screener week prior to randomization.
  Participants
    Yes, one | 20 | 29 | 20 | 69
    Yes, more than one | 15 | 14 | 23 | 52
    No | 92 | 84 | 88 | 264
Chronic Pain [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to affirm or deny chronic pain in different locations of the body (head or face, right hand arm or shoulder, left hand arm or shoulder, right buttock leg or foot, left buttock leg or foot, chest abdomen or pelvis, neck or upper back). These values were combined to determine a total raw score for Chronic Pain. Raw scores range from 0-6, with higher scores indicating chronic pain that's spread out compared to low scores that indicate localized pain.
  units on a scale | 3.0 (2.0) | 2.9 (1.9) | 2.9 (1.9) | 2.9 (1.9)
ITQ score [Mean (Standard Deviation); unit: units on a scale] — The Immersive Tendency Questionnaire is scored by using a scale of 1 (never) to 7 (often) to answer 18 questions that assesses a person's emotional engagement, how often they use digital devices, and how much attention they give to an activity to the point of neglecting their surroundings. Scores can range from 18-126 - higher scores indicate that a person's sense of immersion is intense. ITQ is asked once during the screening week.
  units on a scale | 99.9 (18.1) | 102.2 (17.7) | 99.6 (17.7) | 100.6 (17.7)
Patient Health Questionnaire-2 (PHQ-2) [Mean (Standard Deviation); unit: units on a scale] — PHQ-2 is a two-question screening tool that measures the likelihood of depression. Respondents rate how often they have experienced depressed mood or anhedonia (lack of pleasure in activities) over the past two weeks. Responses to each question are recorded on a Likert scale from 0 to 3, with 0 indicating "not at all" and 3 indicating "nearly every day". A score of 3 or higher indicates a likelihood of major depressive disorder. The total score is the sum of the two responses, ranging from 0 to 6. Questionnaire was sent to participants once during 7-day screening week.
  units on a scale | 1.9 (1.7) | 1.9 (1.8) | 1.7 (1.7) | 1.8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS-PI) at Day 30
Description: The primary outcome for this study will be self-reported pain interference using Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI) version 8a. The pain interference scale measures the consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Items are rated on a 5-point Likert scale from "not at all" (1) to "very much" (5) with a raw score calculated by a sum of the 8 items ranging from 8 to 40. Results are linked to a T-Score (healthmeasures.net) to standardize the results across a general population (a mean T-score of 50 and a standard deviation of 10).
  PROMIS-PI is positively scored, where higher scores indicate worse pain interference. The difference from baseline is reported as Day 30 - baseline, therefore a negative difference corresponds to improvement of symptoms (reduced pain interference).
Time Frame: From baseline to day 30
Population: All analyses will be performed by study arm using an Intent-to-Treat (ITT) population defined as all randomized participants across all three arms. Missing data was accounted for in the overall number of participants analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 108 | 110 | 114
units on a scale | -1.15 (6.63) | -1.86 (5.06) | -1.67 (5.93)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The primary analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS-PI score obtained at Days 7, 15, 21, and 30, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-PI t-score as a continuous covariate; Test type: Other — Primary inference will be based on the treatment comparison of least squares means for Day 30, and a p-value will be presented for this time period only. The null hypothesis is that the mean difference in the primary endpoint between the treatment groups and the sham control group is zero, versus the alternative hypothesis that these differences are not zero; p = 0.4884, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.47, 95% CI 2-sided [-0.87 to 1.81] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8095, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.16, 95% CI 2-sided [-1.12 to 1.43] — Skills-Based VR - Sham VR

2. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS-PI) at Day 60 and Day 90
Description: One of the secondary outcomes for this study will be self-reported pain interference (PI) using Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI) version 8a. The pain interference scale measures the consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Items are rated on a 5-point Likert scale from "not at all" (1) to "very much" (5), with a raw score calculated by a sum of the 8 items ranging from 8 to 40. Results are linked to a T-Score to standardize the results across a general population (a mean T-score of 50 and a standard deviation of 10).
  PROMIS-PI is positively scored, where higher scores indicate worse pain interference. The difference from baseline is reported as Day 60 - baseline and Day 90 - baseline, therefore a negative difference corresponds to improvement of symptoms (reduced PI)
Time Frame: From baseline to day 60, from baseline to end of treatment at day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 127 | 127 | 131
units on a scale
  Day 60 - baseline: number analyzed (Participants) | 103 | 104 | 109
  Day 60 - baseline | -1.32 (6.71) | -2.41 (6.18) | -2.79 (7.73)
  Day 90 - baseline: number analyzed (Participants) | 103 | 106 | 109
  Day 90 - baseline | -1.45 (6.43) | -2.79 (5.23) | -3.51 (7.15)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS-PI score obtained at Days 60 and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-PI t-score as a continuous covariate; Test type: Other — The inference will be based on the treatment comparison of least squares means for Day 60, and a p-value will be presented for this time period only. The null hypothesis is that the mean difference in the primary endpoint between the treatment groups and the sham control group is zero, versus the alternative hypothesis that these differences are not zero; p = 0.3101, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.79, 95% CI 2-sided [-0.74 to 2.32] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.6328, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.42, 95% CI 2-sided [-2.13 to 1.30] — Skills-Based VR - Sham VR
Statistical Analysis 3: Comparison: Distraction-Based VR vs Sham VR; [analysis description as in outcome 2, analysis 1]; Test type: Other — The inference will be based on the treatment comparison of least squares means for Day 90, and a p-value will be presented for this time period only. The null hypothesis is that the mean difference in the primary endpoint between the treatment groups and the sham control group is zero, versus the alternative hypothesis that these differences are not zero; p = 0.1260, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 1.16, 95% CI 2-sided [-0.33 to 2.64] — Distraction-Based VR - Sham VR
Statistical Analysis 4: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 3]; p = 0.5150, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.51, 95% CI 2-sided [-2.05 to 1.03] — Skills-Based VR - Sham VR

3. Secondary Outcome: Change From Baseline in Pain Catastrophizing Survey Short Form 6 (PCS SF-6) at Day 90.
Description: The outcome for this study will be self-reported pain catastrophizing using the Pain Catastrophizing Survey Short Form 6 (PCS SF-6).
  Pain catastrophizing is a negative mental set regarding actual or anticipated pain, and includes aspects of rumination, magnification, and sense of helplessness. PCS is a 6-item short form survey that measures rates of high catastrophizing as defined by a score of ≥7. Items are rated on a 5-point Likert scale from "not at all" (0) to "all the time" (4) with a raw score calculated by a sum of the 6 items ranging from 0 to 24.
  The scale is positively scored, where higher scores indicate greater levels of pain catastrophizing. The difference from baseline is reported as Day 90 - baseline, therefore a negative difference corresponds to improvement of symptoms (reduced pain catastrophizing).
Time Frame: From baseline to end of treatment at day 90
Population: All analyses will be performed by study arm using an Intent-to-Treat (ITT) population defined as all randomized participants. Missing data was accounted for in the overall number of participants analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 103 | 106 | 108
units on a scale | -1.38 (4.69) | -3.04 (4.59) | -3.27 (4.84)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PCS SF-6 score obtained at Days 15, 30, 60, and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PCS SF-6 t-score as a continuous covariate; Test type: Other — Primary inference will be based on the treatment comparison of least squares means for Day 90, and a p-value will be presented for this time period only. The null hypothesis is that the mean difference in the primary endpoint between the treatment groups and the sham control group is zero, versus the alternative hypothesis that these differences are not zero; p = .0180, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 1.43, 95% CI 2-sided [0.25 to 2.61] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.5742, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.33, 95% CI 2-sided [-1.48 to 0.82] — Skills-Based VR - Sham VR

4. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety at Day 90
Description: The primary outcome for this study will be self-reported anxiety using Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety version 4. This scale assesses self-reported perceptions of fear, anxious misery (worry, dread), hyperarousal, and somatic symptoms related to arousal. Items are rated Items are rated on a 5-point Likert scale from "never" (1) to "always" (5), with a raw score calculated by a sum of the 4 items ranging from 4 to 20. Results are linked to a T-Score (healthmeasures.net) to standardize the results across a general population (a mean T-score of 50 and a standard deviation of 10).
  PROMIS-Anxiety is positively scored, where higher scores indicate worse anxiety. The difference from baseline is reported as Day 90 - baseline, therefore a negative difference corresponds to improvement of symptoms (reduced anxiety).
Time Frame: From baseline to end of treatment at day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 102 | 106 | 109
units on a scale | -1.89 (9.14) | -2.88 (9.03) | -1.97 (6.95)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS- Anxiety score obtained at Day 15, 30, 60, and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-Anxiety t-score as a continuous covariate; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.7338, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.39, 95% CI 2-sided [-1.85 to 2.62] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS-Anxiety score obtained at Days 15, 30, 60, and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-Anxiety t-score as a continuous covariate; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.5279, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.63, 95% CI 2-sided [-1.34 to 2.60] — Skills-Based VR - Sham VR

5. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance to Day 90
Description: The secondary outcome for this study will be self-reported Sleep Disturbance using Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance version 6a. This scale assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep.
  Items are rated on a 5-point Likert scale from "not at all" (1) and "very much" (5), with a raw score calculated by a sum of the 6 items ranging from 6 to 30. Results are linked to a T-Score (healthmeasures.net) to standardize the results across a general population (a mean T-score of 50 and a standard deviation of 10).
  PROMIS-Sleep Disturbance is positively scored, where higher scores indicate worse sleep disturbance. The negative difference from baseline corresponds to improvement of symptoms (reduced sleep disturbance).
Time Frame: From baseline to end of treatment at day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 102 | 103 | 109
units on a scale | -2.08 (7.27) | -2.44 (7.14) | -2.76 (7.36)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS-Sleep Disturbance score obtained at Days 15, 30, 60, and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-Sleep Disturbance t-score as a continuous covariate; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.1833, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 1.19, 95% CI 2-sided [-0.56 to 2.94] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 5, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.7006, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.33, 95% CI 2-sided [-2.04 to 1.37] — Skills-Based VR - Sham VR

6. Secondary Outcome: Change From Baseline to Day 90 in Weekly Average Opioid Usage
Description: The secondary outcome for the this study is the change from study baseline to Day 90 in the frequency of self-reported daily opioid use. Participants were asked at baseline and Day 90 "Are you currently taking an opioid pain medication on a daily basis? Yes, No, or Not sure"
  The number of "Yes" responses and the total number of responses is reported.
Time Frame: From baseline to end of treatment at day 90
Population: Responses marked as "Not sure" or missing were excluded from the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 127 | 127 | 131
Participants
  Baseline: number analyzed (Participants) | 125 | 126 | 129
  Baseline | 41 | 36 | 40
  Day 90: number analyzed (Participants) | 101 | 106 | 109
  Day 90 | 26 | 26 | 30
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The Cochran-Mantel-Haenszel (CMH) test was used to compare the association between time (baseline and day 90) and response (yes or no) while stratifying for the treatment groups. The null hypothesis is that the common odds ratio of the association between time and response across the treatment groups is equal to 1, versus the alternative hypothesis that the common odds ratio is not equal to 1; Test type: Other; p = 0.1913, Cochran-Mantel-Haenszel — A two-sided test performed at the 0.05 level of significance without the continuity correction; Common Odds Ratio = 0.76, 95% CI 2-sided [0.50 to 1.15]
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.3670, Cochran-Mantel-Haenszel — A two-sided test performed at the 0.05 level of significance without the continuity correction; Common Odds Ratio = 0.83, 95% CI 2-sided [0.55 to 1.24]

7. Other Pre Specified Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function 6b at Day 90
Description: The exploratory outcome for this study will be self-reported physical function using Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function 6b. The 6-item PROMIS Physical Function scale measures measures self-reported functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living.
  Items are rated on a 5-point Likert scale from "Cannot do" (1) to "Not at all" (5), with a raw score calculated by a sum of the 6 items ranging from 6 to 30.Results are linked to a T-Score (healthmeasures.net) to standardize the results across a general population (a mean T-score of 50 and a standard deviation of 10).
  PROMIS-Physical Function is positively scored, where higher T-scores indicate better physical function. The difference from baseline is reported as Day 90 - baseline, with positive differences indicating better physical function.
Time Frame: From baseline to end of treatment at day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 103 | 106 | 108
units on a scale | 0.74 (4.14) | 1.56 (4.56) | 1.65 (5.16)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS- PF score obtained for Day 15, 30, 60, and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-PF t-score as a continuous covariate; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.1619, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.83, 95% CI 2-sided [-1.98 to 0.33] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.9569, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.04, 95% CI 2-sided [-1.31 to 1.24] — Skills-Based VR - Sham VR

8. Other Pre Specified Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 4 at Day 90
Description: The exploratory outcome for this study will be self-reported depression using Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 4 scale. The 4-item PROMIS Depression scale measures self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Items are rated on a 5-point Likert scale from "never" (1) to "always" (5), with a raw score calculated by a sum of the 4 items ranging from 4 to 20. Results are linked to a T-Score (healthmeasures.net) to standardize the results across a general population (a mean T-score of 50 and a standard deviation of 10).
  PROMIS-PI is positively scored, where higher scores indicate more severe depression. The negative difference from baseline corresponds to improvement of symptoms (reduced depression symptoms).
Time Frame: From baseline to end of treatment at day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 101 | 106 | 108
units on a scale | -2.02 (7.23) | -2.14 (7.37) | -1.60 (7.68)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline PROMIS-Depression score obtained for Day 15, 30, 60, and 90, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline PROMIS-Depression t-score as a continuous covariate; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.9727, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.03, 95% CI 2-sided [-1.80 to 1.86] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 8, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.6427, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 0.43, 95% CI 2-sided [-1.40 to 2.26] — Skills-Based VR - Sham VR

9. Other Pre Specified Outcome: Biometric Data From Fitbit Charge 4 - Change in Average Daily Steps
Description: The change in average daily steps, as measured by FitBit, is an exploratory endpoint to measure the change in daily physical activity of study participants throughout the duration of study participation. For example, higher number of steps across individuals may indicate greater physical activity, and increasing number of steps throughout the study may indicate improving physical activity.
  Data from Fitbit devices were aggregated by Fitabase during a designated window of enrollment. Daily steps were averaged over 7-day periods account for variation in Fitbit adherence, i.e. wearing the device. The average of daily steps taken over the first week of study participation is used as the baseline measurement because Fitbit devices were provisioned to participants after baseline measurements were recorded (e.g. start of treatment). Similarly, an average of daily steps recorded over the final seven days of treatment (to day 90) were measured.
Time Frame: From day 1 to end of treatment at day 90
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 44 | 52 | 46
steps per day | 204.59 (2980.20) | -810.86 (3810.49) | 156.66 (2370.43)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline average weekly steps obtained at weeks 1 thorough 12, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline average weekly steps as a continuous covariate; Test type: Other — The inference will be based on the treatment comparison of least squares means for week 12, and a p-value will be presented for this time period only. The null hypothesis is that the mean difference in the change in the average weekly steps between the treatment groups and the sham control group is zero, versus the alternative hypothesis that these differences are not zero; p = 0.2910, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 691.58, 95% CI 2-sided [-602.98 to 1986.14] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 9, analysis 1]; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.4842, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 405.68, 95% CI 2-sided [-741.79 to 1553.15] — Skills-Based VR - Sham VR

10. Other Pre Specified Outcome: Biometric Data From Fitbit Charge 4 - Change in Average Sleep Score
Description: The change in average sleep score, as measured by FitBit, is an exploratory endpoint to measure the change of sleep quality throughout the duration of study participation. A higher change in sleep score may indicate improvement in the quality of sleep.
  Fitbit calculates sleep score using an algorithm which takes into account heart rate, total time asleep, and stages of sleep. Sleep scores range from 0-100, with the following categories:
  Excellent: 90-100 Good: 80-89 Fair: 60-79 Poor: Less than 60
  The average score ranges from 72 to 83. Data from Fitbit devices were aggregated by Fitabase during a designated window of enrollment. Sleep scores were averaged over 7-day periods account for variation in Fitbit adherence, i.e. wearing the device. The average of sleep scores recorded over the first week of study participation is used as the baseline. Similarly, an average of sleep scores recorded over the final seven days of treatment (to day 90) was measured.
Time Frame: From day 1 to end of treatment at day 90
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 30 | 41 | 31
units on a scale | 0.34 (2.94) | -1.17 (7.69) | -0.61 (3.40)
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; The analysis will compare the treatment groups, separately, to the control group using a linear mixed model repeated measures (MMRM) analysis. The repeated measures are the change from baseline average weekly sleep scores obtained at weeks 1 thorough 12, respectively. The model will include fixed categorical effects for treatment, week, treatment by week interaction, and the baseline sleep score as a continuous covariate; Test type: Other — The inference will be based on the treatment comparison of least squares means for week 12, and a p-value will be presented for this time period only. The null hypothesis is that the mean difference in the change in the average weekly sleep scores between the treatment groups and the sham control group is zero, versus the alternative hypothesis that these differences are not zero; p = 0.4228, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = 1.00, 95% CI 2-sided [-1.48 to 3.49] — Distraction-Based VR - Sham VR
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 10, analysis 1]; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.8363, Mixed Models Analysis — A two-sided test performed at the 0.05 level of significance; Difference in Least Squares Means = -0.28, 95% CI 2-sided [-2.92 to 2.37] — Skills-Based VR - Sham VR

11. Other Pre Specified Outcome: Change in Overall Effect of Treatment From Baseline to Day 90 Measured by Patient's Global Impression of Change (PGIC)
Description: The overall effect of the treatment from study baseline to Day 90, measured by the Patients' Global Impression of Change (PGIC) is an exploratory endpoint to assess the efficacy of Skills-based and Distraction VR. This scale measures self-reported belief regarding efficacy of treatment.
  At Day 90, participants are asked "Since the start of the study, my overall pain is..." with responses on a 7-point Likert scale from "Very much improved" (1) to "Very much worse" (7). Based on the PGIC assessment, a dichotomous scale of "Yes" or "No" was derived. A favorable response of 1-4 on the PGIC indicates "Yes, significant improvement occurred over the course of the study". An unfavorable response of 5-7 indicates "No, significant improvement did not occur over the course of the study".
  Number of participants who scored between 1-4, therefore indicating a significant improvement in their pain levels over the course of the study ("Number of participants with "Yes"), are reported below.
Time Frame: Measured at end of treatment at day 90
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
Number analyzed (Participants) | 103 | 106 | 109
Participants | 53 | 59 | 68
Statistical Analysis 1: Comparison: Distraction-Based VR vs Sham VR; Responder status ("Yes" vs. "No") will be analyzed as the dependent variable using logistic regression, with terms for treatment groups and baseline PROMIS-PI as predictors. The null hypothesis is that there is no difference between the treatment groups, versus the alternative hypothesis that there a difference exists between the treatment groups; Test type: Other; p = 0.514, Regression, Logistic — A two-sided test performed at the 0.05 level of significance; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.48 to 1.44] — Sham VR as the reference group
Statistical Analysis 2: Comparison: Sham VR vs Skills-Based VR; [analysis description as in outcome 11, analysis 1]; Test type: Other; p = 0.280, Regression, Logistic — A two-sided test performed at the 0.05 level of significance; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.78 to 2.36] — Sham VR as the reference group

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during participants' 12-week follow-up period.
Description: Adverse events were collected primarily by a weekly adverse event assessment questionnaire, and events were also reported if participants indicated an adverse event during communications with study team and via other study free-text responses.
  Adverse events were considered moderate if medical intervention, such as use of a medication or an outpatient visit to a medical professional, occurred. Events were considered severe if visits with medical professionals involved an overnight stay.
Arm/Group | Distraction-Based VR | Sham VR | Skills-Based VR
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127 | 0/131
Serious Adverse Events (participants affected / at risk) | 3/127 | 1/127 | 3/131
Other Adverse Events (participants affected / at risk) | 25/127 | 19/127 | 35/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Distraction-Based VR (N=127) | Sham VR (N=127) | Skills-Based VR (N=131)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 — Inpatient hospitalization for cholelithiasis from 12/30/2022 to 1/8/2023 that was unrelated to the intervention. The event was deemed severe, unexpected and was resolved with treatment. The participant discontinued use of the intervention.
Cardiac Arrest and Sepsis (Cardiac disorders) | 1 | 0 | 0 — Cardiac arrest and sepsis from 8/20/2023 to 8/25/2023. Event was unrelated to intervention, unexpected, severe and resolved with treatment. Participant continued to use the intervention.
Unexpected fall and fever (Infections and infestations) | 0 | 1 | 0 — Participant was hospitalized after fall and fever from 5/6/2021 to 5/8/2021. Event was unrelated to intervention, marked as severe, unexpected and resolved with treatment. Participant continued use of intervention.
Hand Infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — Hospitalization due to bacterial infection of the hand from 3/11/2021 to 3/19/2021. Event was unrelated to the intervention, severe, unexpected and resolved with treatment. Participant continued use of the intervention.
Acute-on-chronic Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Participant was hospitalized for intractable, acute-on-chronic low back pain. Event was unrelated to intervention, marked as severe, unexpected and resolved with treatment. Participant continued use of intervention.
Confusion (Psychiatric disorders) | 0 | 0 | 1 — Participant was hospitalized from 3/17/2023 to 3/23/2023. Event was unrelated to intervention, marked as severe, unexpected and resolved with treatment. Participant continued use of intervention.
Cervical fusion (Surgical and medical procedures) | 1 | 0 | 0 — Cervical fusion during the study requiring inpatient rehab hospitalization from 4/17/2023 to 4/27/2023. Event was unrelated to intervention, marked as severe, unexpected and resolved with treatment. Participant continued use of intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Distraction-Based VR (N=127) | Sham VR (N=127) | Skills-Based VR (N=131)
Facial Injury Aggravation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin Allergic Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Blurry Vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Corneal Irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cybersickness (Product Issues) | 1 (2) | 0 (0) | 8 (8)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 8 (13)
Discomfort (Product Issues) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 4 (4) | 2 (2) | 4 (4)
Eye Hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Strain (Eye disorders) | 1 (1) | 3 (4) | 4 (5)
Difficulty Focusing (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Face Pain (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (4) | 5 (6)
Heart Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Flu (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lightheadedness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (2)
Migraines (Nervous system disorders) | 0 (0) | 1 (1) | 1 (6)
Motion Sickness (Ear and labyrinth disorders) | 2 (7) | 0 (0) | 0 (0)
Upper back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial Infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 2 (2) | 1 (2)
Knee Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Survey responses contained 2-week response windows, so responses at a point in time do not necessarily reflect the actual difference in days.

Variation exists in day difference between baseline measurements and start of study intervention due to variation and delays in the shipping of study devices to participants' homes and the availability of participants to complete protocolized onboarding phone calls.

Only 5 of the 7 baseline daily pain scores were required to be randomized into the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT04409353/Prot_001.pdf
  • Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04409353/SAP_003.pdf
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT04409353/ICF_000.pdf